CLINICAL TRIAL: NCT07023809
Title: Exploration of Factors Influencing Chiropractors' Therapeutic Choices in the Management of Aging Patients: an Observational Study
Brief Title: Approaches to Chiropractic Care in Aging Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Isabelle Pagé, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR_IP_Aging_2025
Record Dates: First submitted 2025-06-01; First posted 2025-06-17 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Muskuloskeletal Diseases
Keywords: Aging; manual therapy; safety; chiropractic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chiropractors: All recruited chiropractors will be part of the same participant group. For each chiropractor, we plan to assess between 4 and 10 patients. Our goal is to analyze differences between the "younger" adult population (ages 18 to 49) and the "aging" adult population (ages 50 and older) in the context of care provided by each chiropractor.

SUMMARY:
The goal of this observational study is to understand how chiropractors adjust their therapeutic approaches based on their beliefs, the patient's age, and patient-specific characteristics, with a particular focus on aging patients. The study population includes licensed chiropractors in Quebec treating adult and aging patients in real clinical settings. Patients involved are receiving their usual care and are not the primary focus of the study.

The main questions it aims to answer are:

* How do chiropractors modify their treatment strategies for aging patients?
* What contextual and clinical factors influence these therapeutic decisions?

Researchers will observe chiropractors during routine care to assess treatment characteristics. To do this, participants will:

* Use a sensor to measure the force applied during specific manual treatments.
* Complete brief questionnaires after each treatment to report contextual details.
* Allow for the presence of a researcher during treatment delivery for observational purposes.

Patients will:

* Fill out a short pre-treatment questionnaire.
* Receive their usual care with no interference in the treatment process.
* Be informed in advance and free to decline participation at any point.

This study aims to provide a detailed picture of current chiropractic practices in Quebec related to the care of aging patients, while minimizing disruption to clinical routines.

DETAILED DESCRIPTION:
Chiropractors play a key role in the management of musculoskeletal conditions in aging populations (Hawk et al., 2010). However, due to age-related physiological changes such as decreased bone density and increased tissue fragility, aging patients may face a higher risk of adverse effects from manual therapies-including fractures or hematomas. To ensure patient safety, clinical guidelines recommend adjusting both the selection and intensity of manual interventions for these individuals.

Although chiropractors report adapting their treatments based on age and perceived physical condition, the specific clinical and contextual factors influencing these therapeutic decisions remain poorly understood (Caissy et al., 2024). Perceived patient frailty, body type, and the chiropractor's own clinical experience may all play a role in guiding these choices. Furthermore, while it is assumed that adaptations in technique reflect a reduction in applied force, it is not yet established whether such adjustments result in measurable changes in treatment intensity compared to care provided to younger adults.

This observational study aims to address this gap by examining the factors that influence chiropractors' therapeutic decision-making when delivering manual therapies to both adult and aging patients. In parallel, it will assess whether clinical adaptations are associated with measurable differences in the force applied during treatment.

The primary objective is to identify clinical and contextual factors that influence chiropractors' therapeutic choices, especially when treating patients perceived as frail. The secondary objective is to compare the force applied during manual therapies between two age groups-patients aged 50 and older (aging group) and those aged 18-49 (younger adult group)-to determine if perceived adaptations correspond to actual reductions in applied force.

Hypotheses:

* Chiropractors will adjust their therapeutic choices based on clinical factors indicative of patient frailty, such as age, medical history, physical condition, and clinical presentation.
* The more fragile a patient is perceived to be (evaluated by the Pictorial Fit-Frail Scale and the Clinical Frailty Scale), the more likely the chiropractor will choose techniques considered safer and lower in applied force.
* On average, the force applied during manual therapy will be lower for aging patients compared to younger adults.

Study Design and Procedures:

This study will be conducted in real-world clinical settings in Quebec. The chiropractor is the primary study participant, with the patient acting as a contextual intermediary, receiving their usual care. No modifications to clinical judgment or treatment type will be imposed.

Chiropractors who consent to participate will meet with the lead researcher to review study objectives, data collection procedures, and informed consent procedures. The discussion will help integrate the study into the clinical workflow with minimal disruption. During the data collection day, the chiropractor will treat patients as usual. A researcher will be present to observe the session and place a force sensor beneath the patient if applicable, depending on the treatment type. After each treatment, the chiropractor will complete a short questionnaire (<10 minutes) about the session. At the end of the day, a brief review and clarification session with the researcher (~10 minutes).

Patients will have been informed in advance (via phone, prior visit, or reception staff) that a research project may be taking place during their upcoming visit. On the day of data collection, they will have access to an information sheet and may ask questions before giving informed consent. If they agree, they will receive their usual care, with the presence of a researcher during treatment. A force sensor may be placed under them, depending on the nature of the manual therapy. Participation may add 5-10 minutes to their normal visit duration. Patients will complete a brief 5-question questionnaire either before or after the treatment.

This protocol is designed to minimize disruption to clinical routines. Observing patient care in a natural setting is essential to collecting contextual and force-related data.

The results of this study will provide new insights into clinical reasoning and force modulation during chiropractic care for aging patients. These findings may inform the development of future clinical guidelines aimed at improving both safety and effectiveness of manual therapy in older adults.

Data Analysis : Descriptive statistics will be used to report sample characteristics of both chiropractors and patients. Manual therapy force (measured in Newtons) will be calculated using a MATLAB script developed by the research team, which identifies the peak force manually for each intervention.

To explore the factors influencing chiropractors' therapeutic choices (e.g., spinal manipulation, mobilization, instrument-assisted techniques, use of blocks), a Bayesian statistical approach will be employed. This method allows for the direct estimation of the probability of various predictor effects (e.g., patient age, gender, frailty score, height, weight), while accounting for inter-practitioner variability.

ELIGIBILITY:
Inclusion criteria for chiropractors:

* Be a practicing chiropractor working in a private clinic in Quebec located within approximately 150 km of the Université du Québec à Trois-Rivières.
* Have a patient base mainly composed of younger adults (ages 18 to 49) and aging adults (50 years and older).
* Use diversified manual therapy techniques on the spine and pelvis. This terminology is commonly used in chiropractic and refers to a range of techniques including spinal manipulation, spinal mobilization, instrument-assisted manipulation, and the use of pelvic blocks.

Exclusion criteria for chiropractors:

* Not having a treatment room large enough to accommodate the researcher and her equipment, in addition to the patient.
* Having a schedule that does not allow extending the duration of multiple treatments within a single day.

Inclusion criteria for patients:

* Be an adult aged between 18 and 49 years or 50 years and older.
* Be a regular patient of the chiropractor.

Exclusion criteria for patients:

- New patients, defined as those attending their first or second appointment at the clinic. These visits are typically longer, and it is reasonable to expect that the patient may have more questions during these initial sessions. The presence of a third party could be uncomfortable for a patient who is still adapting to a new type of care or a new chiropractor. We do not wish to interfere with a patient-chiropractor relationship that is still being established.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chiropractors practicing in private clinics in Québec who report treating adult and aging patients presenting with musculoskeletal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Care approaches | From the start of the clinician work day to the end of the clinician work day (1 day)
  The researcher will take handwritten notes of all spinal manual therapies performed by the chiropractors on their patients during the data collection day.

SECONDARY OUTCOMES:
Manual therapy force | From the start of the clinician work day to the end of the clinician work day (1 day)
  For manual therapy delivered by the chiropractor with the patient lying prone and using a posteroanterior vector, a sensor will be placed between the chiropractor's contact point and the patient's skin. The peak force applied will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, DC, MSc, PhD, Principal Investigator — Université du Québec à Trois-Rivières

IPD SHARING:
Plan to Share IPD: Undecided
We plan to use Borealis, the institutional data repository at the university, for storing our IPD. This platform will ensure the long-term preservation of the data, facilitate its discovery, and manage controlled access. Borealis is freely accessible to project staff and offers multiple features to support secure data storage, sharing, and compliance with ethical standards.

REFERENCES:
- [Background] Caissy, D., Brousseau, D., Blanchette, M. A., Grenier, J.-M. & Pagé, I. Étude descriptive de l'expérience des chiropraticiens lors du traitement des patients vieillissants. Mémoire de maîtrise thesis, Montréal ; Trois-Rivières, Université de Montréal ; Université du Québec à Trois-Rivières., (2024).
- [Background] Hawk C, Schneider M, Dougherty P, Gleberzon BJ, Killinger LZ. Best practices recommendations for chiropractic care for older adults: results of a consensus process. J Manipulative Physiol Ther. 2010 Jul-Aug;33(6):464-73. doi: 10.1016/j.jmpt.2010.06.010. PMID 20732584